CLINICAL TRIAL: NCT05733091
Title: Assessment of Functional and Symptom Outcomes for Survivors of Paranasal Sinus, Nasopharyngeal and Skull Base Tumors
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA18-0969; NCI-2023-01436 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Standard of Care — Standard of care assessment of their function including pituitary hormone lab draws, audiogram hearing test, eye exam, teeth and jaw exam (in trismus clinic) and speech and swallowing evaluation

SUMMARY:
To learn about the symptoms and changes our patients experience while receiving treatment for sinonasal or nasopharyngeal cancer

DETAILED DESCRIPTION:
Objectives:

* To estimate the prevalence and severity of adverse and functional outcomes in survivors of benign and malignant paranasal sinus, nasopharynx and skull base tumors.
* To estimate the prevalence of health promotion behaviors during skull base tumor survivorship
* To identify possible mediators or predictors of survivorship outcomes and health behaviors in survivors of skull base tumors.
* To develop a database of demographic, clinicopathologic, recurrence, survival, functional and patient reported outcomes (PROS) for patients with benign and malignant paranasal sinus, nasopharyngeal and skull base tumors.
* To assess the utility and limitations of PROs in evaluating functional impairments and symptom burden in skull base patients.

ELIGIBILITY:
Inclusion criteria:

1. Previously untreated patients with or suspected to have sinonasal malignancy or nasopharyngeal malignancy diagnosis based on either outside pathology report or MD Anderson pathology report.
2. Age ≥ 18 years
3. Plan to obtain the majority of treatment at MDACC including surgery and radiotherapy
4. Ability to understand and willingness to sign written informed consent

Exclusion criteria:

1. History of the previous solid or liquid malignancies, apart from skin cancers treated with local therapy.
2. Existing neurocognitive impairment that is not the result of sinonasal and nasopharyngeal cancers or is treatment.
3. Previous treatment for sinonasal or nasopharyngeal carcinomas, apart from biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
MD Anderson Symptom Inventory Head and Neck Module (MDASI-HN) | through study completion; an average of 1 year
  MD Anderson Symptom Inventory Head and Neck Module (MDASI-HN) is a disease specific PRO instrument validated for patients with head and neck cancer. It is the most commonly utilized instrument in the head and neck cancer population, of which sinonasal and nasopharyngeal tumors are disease subsites.
  Score scale from 0 (symptom has been present) to 10 (the symptom was as bad as you can imagine it could be)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Su, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org